CLINICAL TRIAL: NCT05167851
Title: A Multicentre Two-arm, Phase II Trial Assessing the Safety and Efficacy of First-line Lazertinib and Locally Ablative Radiotherapy in Patients With Synchronous Oligo-metastatic EGFR-mutant Non-small Cell Lung Cancer
Brief Title: The Safety and Efficacy of First-line Lazertinib and Locally Ablative Radiotherapy in Patients With Synchronous Oligo-metastatic EGFR-mutant Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1227
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lazertinib, a combination group of SBRT (Experimental): * Lazertinib 240mg once a day(QD) oral(PO)
    -If there is no disease progression or unacceptable toxicity, treatment is performed at 1 cycle (28 days) interval . This is expected to be an average of one year.
  * Stereotactic Body Radiation Therapy (SBRT) to oligometastatic sites SBRT(Stereotactic Body Radiation Therapy) will be delivered to the primary tumour and to all metastatic sites. SBRT(Stereotactic Body Radiation Therapy) will be delivered using risk-adapted SBRT with a maximum of 5 SBRT(Stereotactic Body Radiation Therapy) fractions.
  Interventions: Drug: Lazertinib , a combination group of SBRT
- Lazertinib single administration group (Active Comparator): * Lazertinib 240mg once a day(QD) oral(PO)
  -If there is no disease progression or unacceptable toxicity, treatment is performed at 1 cycle (28 days) interval . This is expected to be an average of one year.
  Interventions: Drug: Lazertinib single administration group

INTERVENTIONS:
Drug: Lazertinib , a combination group of SBRT — * Lazertinib 240mg once a day(QD) oral(PO)
  -If there is no disease progression or unacceptable toxicity, treatment is performed at 1 cycle (28 days) interval . This is expected to be an average of one year.
  Arms: Lazertinib, a combination group of SBRT
Drug: Lazertinib single administration group — * Lazertinib 240mg once a day(QD) oral(PO)
  -If there is no disease progression or unacceptable toxicity, treatment is performed at 1 cycle (28 days) interval . This is expected to be an average of one year.
  Arms: Lazertinib single administration group

SUMMARY:
This is based on the observations that disease progression under EGFR(Epidermal Growth Factor Receptor) targeting TKI(Tyrosine Kinase Inhibitor) most frequently occurs at the original sites of metastatic disease and that the majority of patients shows disease progression in a limited number of metastatic lesions, a situation defined as oligoprogression.

All studies reported a significantly and clinically relevant improved OS(Overall Survival) or PFS(Period Free Survival) for adding locally ablative therapy to standard of care systemic therapy. However, these studies included only very few NSCLC(non small cell lunc cancer) patients with activating driver mutations and the benefit of adding upfront local radiotherapy might be smaller or larger in this NSCLC(non small cell lunc cancer) patient population with activating driver mutations and treatment with TKIs(Tyrosine Kinase Inhibitor) smaller because of the higher systemic efficacy of TKIs(Tyrosine Kinase Inhibitor) compared to chemotherapy or larger because the benefit of local treatment might become most obvious if potential microscopic disease is successfully controlled by TKI(Tyrosine Kinase Inhibitor)s .Consequently, there is a clinical need to evaluate locally ablative therapy in oligometastatic EGFR (Epidermal Growth Factor Receptor) -mutant NSCLC(non small cell lunc cancer) patients and simultaneously a strong rational that this population might benefit in particular from a combined modality treatment: the benefit of locally ablative therapy is expected to be largest in situations of effective systemic therapies to control locally untreated microscopic disease which is true for EGFR (Epidermal Growth Factor Receptor) targeting.

The investigator therefore propose a prospective two-arm phase II study, which aims to evaluate safety and efficacy of lazertinib combined with early locally ablative radiotherapy of all cancer sites in patients with synchronous oligometastatic (primary tumour and maximum 5 metastases) EGFR (Epidermal Growth Factor Receptor) -mutant (exon 19 deletion or exon 21 L858R) NSCLC. Eradication of all macroscopic cancer sites at the time of primary diagnosis by combined modality treatment is expected to decrease the risk of resistance development with only microscopic disease potentially remaining. This will result in an improvement of PFS(Period Free Survival) and OS(Overall Survival) without added high-grade toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, treatment naïve EGFR-mutant NSCLC, with or without T790M resistance mutation.
2. Presence of the sensitising EGFR-mutation (exon 19 deletion and/or L858R) detected by an accredited laboratory.
3. Synchronous oligometastatic stage IV disease (max 5 lesions)
4. Measurable disease as defined according to RECIST v1.1
5. All lesions amenable for radical radiotherapy according to local judgment
6. Age ≥18 years
7. ECOG performance status 0-2
8. Life expectancy ≥12 months
9. Adequate haematological function:

   * Hemoglobin 90 g/L
   * Absolute neutrophil count (ANC) 1.5× 109/L
   * Platelet count 100× 109/L
10. Adequate renal function:

    Serum creatinine 1.5x ULN or creatinine clearance ≥50 mL/min (calculated according to Cockcroft-Gault, see below). Confirmation of creating clearance is only required when serum creatinine is >1.5x ULN.
11. Adequate liver function:

    * ALT and AST 2.5× ULN. If the patient has liver metastases, ALT and AST must be ≤5× ULN
    * Total serum bilirubin 1.5× ULN. If the patient has documented Gilbert's syndrome (unconjugated hyperbilirubinaemia) 3× ULN.
12. Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 7 days before enrolment.
13. Written IC for protocol treatment must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

1. Prior chemotherapy, immunotherapy, radiotherapy or therapeutical surgery for NSCLC (an exception is the resection of CNS or adrenal metastases)
2. More than 5 distant oligometastases (any second intra-thoracic lesion will count as a distant metastasis; regional nodal metastases will not count to the 5 oligometastases) and more than 2 intra-thoracic lesions.
3. Brain metastases not amenable for radiosurgery or neurosurgery
4. Presence of leptomeningeal metastases
5. Symptomatic spinal cord compression
6. Extracranial metastatic locations such as malignant ascites, pleural or pericardial effusion, diffuse lymphangiosis of skin or lung, diffuse bone marrow metastasis, abdominal masses/abdominal organomegaly, identified by physical exam that is not measurable by reproducible imaging techniques.
7. Currently receiving (or unable to stop use prior to receiving the first dose of lazertinib treatment) medications or herbal supplements known to be potent CYP3A4 inducers that cannot be stopped before enrolment and for the duration of the trial.
8. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol.

   Patients with a resolved or chronic HBV infection are eligible if they are:
   * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG] or
   * Positive for HBsAg, negative for HBeAg but for >6 months have had transaminases levels below ULN and HBV DNA levels below 2000 IU/mL (i.e., are in an inactive carrier state).
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of lazertinib
10. Any of the following cardiac criteria:

    QTcF >470 msec obtained from 3 ECGs, using the screening clinic ECG machine derived QTc value (QTcF: corrected QT interval using Fredericia's formula).

    Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block or second degree heart block).

    Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes (TdP).
11. Past medical history of ILD, drug induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
12. Idiopathic pulmonary fibrosis which is a contraindication to lung radiation.
13. History of hypersensitivity to active or inactive excipients of lazertinib or drugs with a similar chemical structure or class to lazertinib.
14. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements Women who are pregnant or in the period of lactation.
15. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method (Please refer to 8.4 for highly effective contraceptive methods) during the trial and up to 6 weeks for women and up to 4 months for men, after discontinuing lazertinib treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | every 8 weeks after enrollment, an average of one year
  The time to recurrence/progression/death and From start of Lazertinib to documented radiographic relapse/progression by RECIST 1.1 criteria
Progression free survival (PFS) | disease progression, an average of one year
  The time to recurrence/progression/death and From start of Lazertinib to documented radiographic relapse/progression by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | Every 12 weeks after the end of the study , which will be conducted in about 3 years.
  Overall survival (OS) is defined as the time from the date of enrolment until death from any cause. Censoring will occur at the last follow-up date.
Distant Progression free survival (Distant PFS) | At screening, every 8 weeks after enrollment, and when the disease progresses. This is expected to be an average of one year.
  Distant PFS is defined as the time from date of enrollment until development of new metastases, excluding oligometastases diagnosed at enrolment.
Objective response rate (ORR) | At screening, every 8 weeks after enrollment, and when the disease progresses. This is expected to be an average of one year.
  Objective response rate (ORR) is defined as the percentage of patients that achieve a best overall response [complete response (CR) or partial response (PR)] according to RECIST v1.1 from enrolment across all trial assessment time-points.
Duration of Response (DoR) | At screening, every 8 weeks after enrollment, and when the disease progresses. This is expected to be an average of one year.
  Duration of Response (DoR) is defined as the interval from the date of first documentation of objective response (CR or PR, according to RECIST v1.1) to the date of first documented progression, relapse or death.
Adverse event according to CTCAE(Common Terminology Criteria for Adverse Event) v5.0 | Screening, every cycle visit and End of study, and evaluation up to 6 weeks after End of the study. This is is expected to be an average of one year.
  AE captured by CYCAE 5.0 until after 30days of last administration.
Pattern of disease progression | At screening, every 8 weeks after enrollment, and when the disease progresses. This is expected to be an average of one year.
  The pattern of disease progression is defined as the site of first progression: None, locoregional, distant (bone, brain, liver, etc) or both locoregional and distant, evaluated up to 18-months post enrollment.
Exploratory analysis (Analysis of acquired resistance mechanism through cfDNA) | At Screening and disease progression. This is expected to be an average of one year.
  • Analysis of acquired resistance mechanisms to lazertinib plus radiotherapy at the time of progression using tumor/liquid cfDNA biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Sun min Lim, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu CY, Hsia TC, Lin YC, Liang JA, Li CC, Chien CR. Efficacy of Definitive Radiotherapy for Patients with Clinical Stage IIIB or IIIC Lung Adenocarcinoma and Epidermal Growth Factor Receptor (EGFR) Mutations Treated Using First- or Second-Generation EGFR Tyrosine Kinase Inhibitors. Can Respir J. 2024 Mar 5;2024:8889536. doi: 10.1155/2024/8889536. eCollection 2024. PMID 38476120
- [Derived] Kim KH, Yoon S, Ahn HK, Lee SY, Lee GW, Lee SS, Cho JH, Cho BC, Yoon HI, Lim SM. A Multicenter Two-arm, Phase II Trial Assessing the Safety and Efficacy of First-line Lazertinib and Locally Ablative Radiotherapy in Patients With Synchronous Oligo-metastatic EGFR-mutant Non-small Cell Lung Cancer (ABLATE, KCSG-LU21-11). Clin Lung Cancer. 2022 Dec;23(8):e536-e539. doi: 10.1016/j.cllc.2022.07.014. Epub 2022 Aug 7. PMID 36002368